CLINICAL TRIAL: NCT02690467
Title: Efficacy, Safety and Acceptability of the New Pen Needle 33G x 4 mm: a Cross-over Randomised Non Inferiority Trial
Brief Title: Efficacy, Safety and Acceptability of the New Pen Needle 34gx3,5mm.
Acronym: AGO 02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Outcomes Research and Clinical Epidemiology, Italy (Other)
Collaborators: Artsana S.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGO 02
Record Dates: First submitted 2016-02-02; First posted 2016-02-24 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
Keywords: Insulin therapy; Needle
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insupen G34x3,5mm (Experimental): Needle for insulin pen 3,5 mm long and with a diameter of 34 gauge
  Interventions: Device: Insupen G34x3,5mm
- Insupen G32x4mm (Active Comparator): Needle for insulin pen 4 mm long and with a diameter of 32 gauge
  Interventions: Device: Insupen G32x4mm

INTERVENTIONS:
Device: Insupen G34x3,5mm
  Arms: Insupen G34x3,5mm
Device: Insupen G32x4mm
  Arms: Insupen G32x4mm

SUMMARY:
The purpose of this study is to determine the non-inferiority of a new Pic Insupen 34Gx3,5mm needle vs. a 32Gx4mm needle in terms of metabolic control, safety and acceptability in patients with diabetes treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Age >= 18 years
* Multiple daily injections of insulin for at least 6 months
* Signed informed consent

Exclusion Criteria:

* Pregnancy or or breast feeding
* Inability to fill in the questionnaire
* Combined therapy for diabetes (oral drugs associated with insulin injections)
* Any medical condition that could interfere with the study according to the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
Fructosamine levels | 3 weeks
  Change from baseline in fructosamine levels after 3 weeks of treatment

SECONDARY OUTCOMES:
Glycemic variability expressed as the standard deviation of fasting blood and postprandial glucose levels | 3 weeks
  Change from baseline in glycemic variability after 3 weeks of treatment
Daily insulin dose | 3 weeks
  Change from baseline in daily insulin dose after 3 weeks of treatment
Body weight | 3 weeks
  Change from baseline in body weight after 3 weeks of treatment
Pain | 3 weeks
  Pain measured by visual analogue scale after 3 weeks of treatment
Patient satisfaction measured by a questionnaire | 3 weeks
  Patient satisfaction measured by a questionnaire after 3 weeks of treatment
Number of patients with hypoglycaemia | 3 weeks
  Number of patients with hypoglycaemia during 3 weeks
Number of hypoglycaemia episodes | 3 weeks
  Total number of phypoglycaemia episodes during 3 weeks
Number of episodes of insulin leakage at injection site | 3 weeks
  Number of episodes of insulin leakage at injection site during 3 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - U.O. Malattie Metaboliche e Diabetologia - Ospedale Treviglio, Treviglio, BG
  - Struttura Semplice Dipartimentale di Diabetologia e Malattie Metaboliche - Az. Osp. S. Anna - PO Cantù, Mariano Comense, CO
  - Struttura Semplice Dipartimentale Diabetologia, Endocrinologia e Nutrizione Clinica - Az. Osp. Desio e Vimercate, Desio, MI
  - Struttura Complessa Dietologia - Diabetologia Malattie Metaboliche - Ospedale Pertini, Roma, RM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Berardis G, Scardapane M, Lucisano G, Abbruzzese S, Bossi AC, Cipponeri E, D'Angelo P, Fontana L, Lancione R, Marelli G, Sciangula L, Nicolucci A. Efficacy, safety and acceptability of the new pen needle 34G x 3.5 mm: a crossover randomized non-inferiority trial; AGO 02 study. Curr Med Res Opin. 2018 Sep;34(9):1699-1704. doi: 10.1080/03007995.2018.1491396. Epub 2018 Jul 5. PMID 29924641